CLINICAL TRIAL: NCT01074970
Title: PARP Inhibition After Preoperative Chemotherapy in Patients With Triple Negative Breast Cancer or ER/PR +, HER2 Negative With Known BRCA1/2 Mutations: Hoosier Oncology Group BRE09-146
Brief Title: PARP Inhibition for Triple Negative Breast Cancer (ER-/PR-/HER2-)With BRCA1/2 Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRE09-146
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: PARP inhibition + breast cancer; breast cancer; PARP inhibitor; Triple negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Cisplatin Monotherapy (Active Comparator): Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Interventions: Drug: Cisplatin
- Arm B: Combination Therapy (Active Comparator): Rucaparib 24mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
  Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Interventions: Drug: Rucaparib; Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Arms: Arm A: Cisplatin Monotherapy
Drug: Rucaparib — Rucaparib 24mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
  Arms: Arm B: Combination Therapy
Drug: Cisplatin — Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Arms: Arm B: Combination Therapy

SUMMARY:
The purpose of this trial is to evaluate 2-year disease-free survival in this patient population treated with single agent cisplatin and patients treated with cisplatin in combination with Rucaparib following preoperative chemotherapy. Side effects and tolerability of this treatment in patients with residual disease following preoperative chemotherapy will also be observed and characterized.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Safety Run-in will be for the first 12 patients on study only (6 in cohort 1 and 6 in cohort 2). Patients in the safety run will be included in the efficacy analysis on intent to treat basis:

Cisplatin 75 mg/m2 IV D1 every 3 weeks x 4 cycles; Rucaparib 16-30 mg IV D 1,2,3 every 3 weeks x 4 cycles

If cycle 1 is well tolerated, the dose of Rucaparib will be escalated from 16 mg to 24 mg for subsequent cycles in the cohort 1, and 24 mg to 30 mg in the cohort 2.

If ≤ 1 of 6 patients in cohort 1 experiences DLT, cohort 2 will commence. If 2 or more of 6 patients in cohort 1 experience DLT, the study will be suspended and an amendment to explore lower doses will be considered.

If ≤ 1 of 6 patients in cohort 2 experiences DLT, the randomized portion of the study will commence. If 2 or more of 6 patients experience DLT, the study will be suspended and an amendment to proceed with the randomized portion at the cohort 2 dose (24 mg) will be considered.

During the randomized portion of the study, patients will be randomized to either Arm A or Arm B.

Stratification factors:

* Anthracycline vs. not
* Residual LN involvement vs. No Residual LN involvement

Arm A (Cisplatin Monotherapy) Cisplatin 75 mg/m2 IV D1 every 3 weeks x 4 cycles

Arm B (Combination Therapy) Cisplatin 75 mg/m2 IV D1 every 3 weeks x 4 cycles; Rucaparib 16-30 mg IV D1,2,3 every 3 weeks x 4 cycles

Rucaparib maintenance 30 mg IV weekly x 24 weeks

ECOG Performance Status 0-1

Life Expectancy: Not Specified

Hematopoietic:

* Hemoglobin (Hgb) > 9.0 g/dL
* Platelets > 100 K/ mm3
* Absolute neutrophil count (ANC) > 1.5 K/mm3

Hepatic:

* Bilirubin < upper limit of normal (except in patients with documented Gilbert's disease, who must have a total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST, SGOT) < 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) < 2.5 x ULN

Renal:

* Calculated creatinine clearance of > 50 cc/min using the Cockcroft-Gault formula

Cardiovascular:

* Left ventricular ejection fraction within normal limits.
* Patients with an unstable angina or myocardial infarction within 12 months of study entry are excluded.
* No clinically significant arrhythmia or baseline ECG abnormalities in the opinion of the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed triple negative (ER-/PR-/HER2-) invasive breast cancer, stage I-III at diagnosis (AJCC 6th edition) based on initial evaluation by clinical examination and/or breast imaging. NOTE: Patients with ER+ and/or PR+ may enroll ONLY if they are known carriers of a deleterious mutation in BRCA1 or BRCA2. Patients with HER2+ tumors may not enroll regardless of BRCA status.
* Must have completed preoperative (neoadjuvant) chemotherapy. NOTE: Acceptable preoperative regimens include an anthracycline or a taxane, or both. Patients may NOT have received cisplatin as part of their neoadjuvant therapy regimen. Patients who received preoperative therapy as part of a clinical trial may enroll. No adjuvant chemotherapy after surgery other than that specified in this protocol is allowed. Adjuvant bisphosphonate use is allowed.
* Must have completed definitive resection of primary tumor. The last surgery for breast cancer must have been completed at least 14 days prior to registration for protocol therapy.
* Must have significant residual invasive disease at the time of definitive surgery following preoperative chemotherapy. Significant residual disease is defined at least one of the following:

  * Miller-Payne response in the breast of 0-25.
  * Residual Cancer Burden (RBC) classification II or III6
  * Residual carcinoma in one or more regional lymph nodes that would meet AJCC 6th edition criteria for N1 - N3 disease.
  * Alternatively, if Miller-Payne or RCB grading is not available, the patient will be eligible if the pathology report indicates that the area of residual invasive disease in the breast measures at least 2 cm following preoperative therapy. The presence of DCIS without invasion does not qualify as residual disease in the breast.
* Whole breast radiotherapy is required for patients who underwent breast conserving therapy, including lumpectomy or partial mastectomy. Patients receiving adjuvant radiation therapy must have completed radiotherapy at least 14 days prior to registration for protocol therapy.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Must consent to allow submission of archived tumor tissue sample from definitive surgery.
* Must consent to collection of blood samples for PK analysis.
* Women of childbearing potential and males must be willing to use an effective method of contraception from the time consent is signed until 4 weeks after treatment discontinuation.
* Women of childbearing potential must have a negative pregnancy test within 14 days prior to registration for protocol therapy.
* Women must not be breastfeeding.

Exclusion Criteria:

* No stage IV (metastatic) disease, however no specific staging studies are required in the absence of symptoms or physical exam findings that would suggest distant disease.
* No treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* No history of chronic hepatitis B or C
* No clinically significant infections as judged by the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-02; Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D. Miller, M.D., Study Chair — Hoosier Cancer Research Network
Locations (27):
- United States (27):
  - St. Jude Heritage Healthcare, Fullerton, California
  - University of California Los Angeles, Los Angeles, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Memorial Cancer Institute Breast Cancer Center, Hollywood, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Inc./IU Health Arnett, Lafayette, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Metro Health Cancer Care, Wyoming, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The Center for Cancer & Hematologic Disease, Cherry Hill, New Jersey
  - Virtua Health Cancer Program, Mount Holly, New Jersey
  - South Jersey Health Care, Vineland, New Jersey
  - Presbyterian Medical Group, Albuquerque, New Mexico
  - University of New Mexico Cancer Center: Albuquerque, Albuquerque, New Mexico
  - HOPE a Women's Cancer Center, Asheville, North Carolina
  - Seidman Cancer Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Pinnacle Health Fox Chase Regional Cancer Center, Harrisburg, Pennsylvania
  - Bux-Mont Oncology Hematology Associates (FCCC) at Grand View Hospital, Sellersville, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Background] S. R. Malireddy, S. M. Perkins, S. S. Badve, G. W. Sledge, K. Miller. PARP inhibition after preoperative chemotherapy in patients with triple negative breast cancer (TNBC) or known BRCA1/2 mutations: Hoosier oncology group BRE09-146. J Clin Oncol 29: 2011 (suppl; abstr TPS130)
- [Background] S. Dwadasi, Y. Tong, T. Walsh, M.A. Danso, C.X. Ma, P.A Silverman, M.C. King, S.M. Perkins, S.S. Badve, K. Miller. Cisplatin with or without rucaparib after preoperative chemotherapy in patients with triple negative breast cancer: Hoosier Oncology Group BRE09-146. J Clin Oncol 32:5s, 2014 (suppl; abstr 1019^)
- [Result] Miller K, Tong Y, Jones DR, Walsh T, Danso MA, Ma CX, Silverman P, King MC, Badve SS, Perkins SM. Cisplatin with or without rucaparib after preoperative chemotherapy in patients with triple negative breast cancer: Final efficacy results of Hoosier Oncology Group BRE09-146. J Clin Oncol 33:5s, 2015 (suppl; abstr 1082)
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Cohort 1: Rucaparib 24 mg With Cisplatin: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
  Rucaparib: 24 mg of Rucaparib will be administered on day 1-3 of every 21 days for cycle 2-4 via IV infusion followed in one hour by Cisplatin.
- Safety Cohort 2: Rucaparib 30 mg With Cisplatin: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
  Rucaparib: 30 mg of Rucaparib will be administered on day 1-3 of every 21 days for cycle 2-4 via IV infusion followed in one hour by Cisplatin.
- Arm A: Cisplatin Monotherapy: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
- Arm B: Combination Therapy: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
  Rucaparib: Rucaparib dose should be increased to 30 mg day 1-3 of every 21 days for cycles 2-4 in the absence of dose limiting toxicity in cycle 1.
Period: Overall Study
Arm/Group | Safety Cohort 1: Rucaparib 24 mg With Cisplatin | Safety Cohort 2: Rucaparib 30 mg With Cisplatin | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy
Started | 7 | 6 | 65 | 57
Completed | 3 | 5 | 44 | 40
Not Completed | 4 | 1 | 21 | 17
Not completed — Never Treated | 0 | 0 | 8 | 1
Not completed — Adverse Event | 1 | 0 | 4 | 3
Not completed — Disease progression during treatment | 3 | 1 | 2 | 9
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm B: Combination Therapy; Safety Cohort 2: Rucaparib 30 mg With Cisplatin: Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Rucaparib 24mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
- Safety Cohort 1: Rucaparib 24 mg With Cisplatin: Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Rucaparib 16mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
- Total: Total of all reporting groups
Arm/Group | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy | Safety Cohort 1: Rucaparib 24 mg With Cisplatin | Safety Cohort 2: Rucaparib 30 mg With Cisplatin | Total
Number analyzed (Participants) | 65 | 57 | 7 | 6 | 135
Age, Continuous [Median (Full Range); unit: years] | 48 [27 to 69] | 47 [25 to 75] | 46 [29 to 56] | 49 [21 to 56] | 47 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 57 | 7 | 6 | 135
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 0 | 0 | 9
  Not Hispanic or Latino | 57 | 48 | 7 | 5 | 117
  Unknown or Not Reported | 2 | 6 | 0 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 2 | 1 | 26
  White | 49 | 41 | 5 | 5 | 100
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 65 | 57 | 7 | 6 | 135
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead
  Participants
    ECOG PS 0 | 52 | 49 | 0 | 3 | 104
    ECOG PS 1 | 13 | 8 | 0 | 3 | 24
    Not Collected or Available | 0 | 0 | 7 | 0 | 7
BRCA2 Status Known at Entry [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 0 | 0 | 4
  No | 63 | 55 | 7 | 6 | 131

OUTCOME MEASURES:

1. Primary Outcome: Two-year Disease Free Survival
Description: To evaluate 2-year disease-free survival (DFS), in patients with confirmed TNBC or ER/PR + HER2-, known BRCA1/2 mutations treated with single agent cisplatin and patients treated with cisplatin in combination with Rucaparib following preoperative chemotherapy
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B: Combination Therapy: Rucaparib 24mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
  Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
  Rucaparib: Rucaparib 24mg C1,30mg C2-4, D1,2,3 every 21 days for 4 cycles
  Cisplatin: Cisplatin 75 mg/m2 IV infusion over 60 minutes, D1 every 21 days for 4 cycles
Arm/Group | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy
Number analyzed (Participants) | 65 | 63
percentage of participants | 54.2 [39.8 to 66.6] | 64.1 [50.3 to 75.0]

2. Secondary Outcome: Five-year Disease Free Survival
Description: To evaluate 5-year DFS, in patients with confirmed TNBC or ER/PR + HER2-, known BRCA1/2 mutations treated with single agent cisplatin and patients treated with cisplatin in combination with Rucaparib following preoperative chemotherapy
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy
Number analyzed (Participants) | 65 | 63
percentage of participants | 38.3 [24.6 to 51.8] | 50.1 [35.5 to 63.0]

3. Secondary Outcome: Overall Survival
Description: To determine 5-year overall survival
Time Frame: 60 months
Population: Data for this secondary objective was not collected or analyzed
Arm/Group | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Summarize Grade 2,3, # 4 Toxicities
Description: To characterize the side effects and tolerability of cisplatin and cisplatin plus Rucaparib in patients with residual disease following preoperative chemotherapy by summarizing Grade 2,3, # 4 toxicities according to CTCAE v3.0
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Arm A: Cisplatin Monotherapy | Arm B: Combination Therapy
Number analyzed (Participants) | 65 | 63
participants
  Neutropenia Gr 2 | 16 | 13
  Neutropenia Gr 3 | 11 | 16
  Neutropenia Gr 4 | 0 | 1
  Neutropenic fever Gr 2 | 1 | 1
  Anemia Gr 2 | 5 | 7
  Thrombocytopenia Gr 2 | 2 | 0
  Thrombocytopenia Gr 3 | 0 | 2
  Nausea Gr 2 | 13 | 16
  Nausea Gr 3 | 0 | 3
  Anorexia Gr 2 | 3 | 7
  Fatigue Gr 2 | 14 | 11
  Fatigue Gr 3 | 3 | 6
  Fatigue Gr 4 | 1 | 0
  Tinnitus Gr 2 | 16 | 12
  Tinnitus Gr 3 | 1 | 1
  Nephropathy Gr 2 | 1 | 2
  Neuropathy Gr 2 | 1 | 3
  Neuropathy Gr 3 | 0 | 1
  Vomiting Gr 2 | 5 | 7
  Vomiting Gr 3 | 0 | 3
  Hepatic abnormality Gr 3 | 1 | 3
  Hepatic abnormality Gr 4 | 1 | 0
  Rash Gr 2 | 2 | 2
  Headache Gr 2 | 2 | 5
  Dysguesia Gr 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Arm A : Cisplatin Monotherapy: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
- Arm B : Combination Therapy: Cisplatin: 75 mg/m^2 of Cisplatin will be administered via IV infusion over 60 minutes on day 1 of every 21 days for 4 cycles.
  Rucaparib: 24 mg of Rucaparib will be administered on day 1-3 of every 21 days for cycle 1 via IV infusion followed in one hour by Cisplatin. Rucaparib dose should be increased to 30 mg day 1-3 of every 21 days for cycles 2-4 in the absence of dose limiting toxicity in cycle 1.
Arm/Group | Arm A : Cisplatin Monotherapy | Arm B : Combination Therapy | Safety Cohort 1: Rucaparib 24 mg With Cisplatin
All-Cause Mortality (participants affected / at risk) | 26/66 | 25/63 | 5/7
Serious Adverse Events (participants affected / at risk) | 1/65 | 6/63 | 1/7
Other Adverse Events (participants affected / at risk) | 56/65 | 61/63 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A : Cisplatin Monotherapy (N=65) | Arm B : Combination Therapy (N=63) | Safety Cohort 1: Rucaparib 24 mg With Cisplatin (N=7)
SECONDARY MALIGNANCY - POSSIBLY RELATED TO CANCER TREATMENT (SPECIFY, __) (General disorders) | 1 (1) | 0 (0) | 0 (0)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 0 (0) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MOOD ALTERATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
PAIN (General disorders) | 0 (0) | 2 (2) | 0 (0)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A : Cisplatin Monotherapy (N=65) | Arm B : Combination Therapy (N=63) | Safety Cohort 1: Rucaparib 24 mg With Cisplatin (N=7)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 1 (1) | 4 (10) | 0 (0)
ALKALINE PHOSPHATASE (Investigations) | 5 (5) | 6 (9) | 0 (0)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
ALLERGY/IMMUNOLOGY (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 2 (4) | 5 (7) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 14 (17) | 12 (26) | 5 (20)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 2 (5) | 6 (7) | 0 (0)
AUDITORY/EAR (Ear and labyrinth disorders) | 1 (1) | 6 (6) | 0 (0)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1) | 1 (1) | 0 (0)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 20 (27) | 28 (40) | 4 (8)
CONSTITUTIONAL SYMPTOMS (General disorders) | 5 (5) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (8) | 5 (5)
CREATININE (Investigations) | 2 (2) | 4 (11) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 8 (14) | 2 (2)
DENTAL: TEETH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DERMAL CHANGE LYMPHEDEMA, PHLEBOLYMPHEDEMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 4 (8) | 10 (13) | 1 (1)
DIZZINESS (Nervous system disorders) | 3 (3) | 10 (12) | 0 (0)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (8) | 1 (1)
EDEMA: LIMB (General disorders) | 8 (9) | 13 (15) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 33 (56) | 37 (137) | 5 (21)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (2) | 3 (3) | 1 (1)
FLU-LIKE SYNDROME (General disorders) | 1 (1) | 1 (1) | 0 (0)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Metabolism and nutrition disorders) | 7 (15) | 9 (18) | 0 (0)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 3 (3)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 6 (6) | 8 (9) | 3 (6)
HEMOGLOBIN (Blood and lymphatic system disorders) | 17 (21) | 21 (32) | 1 (5)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
HOT FLASHES/FLUSHES (Vascular disorders) | 3 (3) | 4 (9) | 1 (2)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1) | 5 (5) | 2 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS (Infections and infestations) | 8 (9) | 7 (8) | 2 (2)
INFECTION WITH UNKNOWN ANC (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
INSOMNIA (Psychiatric disorders) | 5 (5) | 13 (15) | 4 (9)
LEUKOCYTES (TOTAL WBC) (Investigations) | 13 (28) | 17 (53) | 0 (0)
LYMPHATICS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LYMPHEDEMA-RELATED FIBROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
LYMPHOPENIA (Investigations) | 7 (14) | 13 (22) | 0 (0)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 0 (0)
METABOLIC/LABORATORY (Investigations) | 1 (2) | 0 (0) | 0 (0)
MOOD ALTERATION (Psychiatric disorders) | 12 (14) | 8 (13) | 3 (7)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) (Gastrointestinal disorders) | 5 (5) | 7 (7) | 1 (2)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) (Gastrointestinal disorders) | 2 (2) | 4 (6) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 0 (0)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 0 (0)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 44 (63) | 45 (90) | 7 (21)
NEUROLOGY (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
NEUROPATHY: SENSORY (Nervous system disorders) | 11 (13) | 17 (27) | 3 (5)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 33 (69) | 36 (89) | 4 (6)
OCULAR/VISUAL (Eye disorders) | 3 (4) | 1 (1) | 0 (0)
OTITIS, MIDDLE EAR (NON-INFECTIOUS) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 28 (47) | 44 (129) | 5 (19)
PAIN - OTHER (General disorders) | 8 (9) | 12 (14) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
PLATELETS (Investigations) | 4 (6) | 6 (11) | 2 (2)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 3 (3) | 7 (13) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 0 (0)
PSYCHOSIS (HALLUCINATIONS/DELUSIONS) (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (4) | 0 (0)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0)
RENAL/GENITOURINARY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
SWEATING (DIAPHORESIS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
TASTE ALTERATION (DYSGEUSIA) (Nervous system disorders) | 7 (11) | 4 (4) | 3 (5)
TINNITUS (Ear and labyrinth disorders) | 17 (23) | 17 (32) | 1 (1)
TRISMUS (DIFFICULTY, RESTRICTION OR PAIN WHEN OPENING MOUTH) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
VISION-BLURRED VISION (Eye disorders) | 2 (3) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 10 (12) | 20 (43) | 1 (1)
WEIGHT GAIN (Investigations) | 1 (1) | 1 (2) | 0 (0)
WEIGHT LOSS (Investigations) | 2 (2) | 0 (0) | 0 (0)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
BLOOD/BONE MARROW (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CERVICAL SPINE-RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DRY EYE SYNDROME (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
EDEMA: HEAD AND NECK (General disorders) | 0 (0) | 1 (1) | 0 (0)
EDEMA: TRUNK/GENITAL (General disorders) | 0 (0) | 3 (5) | 0 (0)
EDEMA: VISCERA (General disorders) | 0 (0) | 1 (1) | 0 (0)
ENTERITIS (INFLAMMATION OF THE SMALL BOWEL) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
EXTREMITY-LOWER (GAIT/WALKING) (General disorders) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 4 (6) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
GLOMERULAR FILTRATION RATE (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
HEMORRHAGE, GU (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
INCONTINENCE, URINARY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
INTRA-OPERATIVE INJURY (General disorders) | 0 (0) | 1 (1) | 0 (0)
MAGNESIUM, SERUM-HIGH (HYPERMAGNESEMIA) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY: CRANIAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY: MOTOR (Nervous system disorders) | 0 (0) | 6 (7) | 0 (0)
OPHTHALMOPLEGIA/DIPLOPIA (DOUBLE VISION) (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
PHLEBOLYMPHATIC CORDING (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
RIGORS/CHILLS (General disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (FAINTING) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
VIRAL HEPATITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHAGE, GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
JOINT-FUNCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
UVEITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-09-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT01074970/Prot_SAP_000.pdf